CLINICAL TRIAL: NCT02096068
Title: Neuroprotection With Dexmedetomidine in Patients Undergoing Elective Cardiac or Abdominal Surgery (NEUPRODEX)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Claudia Spies (Other)
Responsible Party: Sponsor-Investigator, Claudia Spies, Department of Anesthesiology and Intensive Care Medicine CVK/CCM, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Neuprodex
Record Dates: First submitted 2014-03-21; First posted 2014-03-26 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Delirium; Postoperative Cognitive Deficit (POCD)
Keywords: Neuroprotection
MeSH Terms: conditions — Delirium | interventions — Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Study group (Experimental): Application of Dexmedetomidine (Dexdor®) perioperatively for a maximum of 48 hours
  Dosing Scheme:
  during operation and mechanical ventilation: 0,7μg/kgABW/h; recovery time until extubation: 0,4μg/kgABW/h; after extubation: 0,2-1,4μg/kgABW/h
  Interventions: Drug: Dexmedetomidine (Dexdor®)
- Control group (Placebo Comparator): Application of placebo for a maximum of 48 hours
  Interventions: Drug: 0.9% Sodium Chloride
- POCD control group (No Intervention): A non-surgical control group of 15 ASA II/III- patients is collected for measuring the learning experience during the cognitive testings. The participants are matched on age, education, and gender to the study patients.

INTERVENTIONS:
Drug: Dexmedetomidine (Dexdor®) — Dexmedetomidine (Dexdor 100 micrograms/ml concentrate for solution for infusion)
  Arms: Study group
Drug: 0.9% Sodium Chloride — Solution for infusion: Sodium Chloride : 9.0 g/l; Each ml contains 9 mg sodium chloride mmol/l : Na+ : 154. Cl-: 154.
  Arms: Control group

SUMMARY:
The drug Dexmedetomidine will be investigated in 72 patients (men and women) undergoing elective cardiac or abdominal surgery. The study medication will be administered perioperatively by intravenous infusion continuously (at the longest 48 h) to prevent/reduce the rate of Delirium and the incidence of postoperative cognitive deficit (POCD).

A non-surgical control group of 15 ASA II/III- patients from Berlin and surrounding area is collected for measuring the learning experience during the cognitive testings. The participants are matched on age, education, and gender to the study patients.

Cognitive testings are performed in patients of the study group (n= 72) and the control group (n= 15) to evaluate deficits in their cognitive areas (POCD (Postoperative cognitive deficit)) at three different time points up to three months.

ELIGIBILITY:
Study Group:

Inclusion Criteria:

1. Patients aged ≥ 60 years
2. Male and female patients undergoing elective cardiac (elective CABG-surgery without valve surgery with left ventricular ejection fraction ≥ 30%) or pancreatic or hepatic or gastric or intestinal surgery of both Campus Charité Mitte and Campus Virchow - Klinikum, Charité - Universitätsmedizin Berlin
3. Offered patient information and written consent by the patient (according to German Drug Law § 40 (1) 3b)
4. Premedication only with benzodiazepines
5. Pain therapy during the operation with regional procedures and/or Sufentanil/Fentanyl
6. Anesthesia in cardio surgery according to Heart-Lung-Apparatus
7. Anesthesia with hypnotic agent Propofol
8. Pain therapy after operation according to S3-Guideline
9. Postoperative medication for anxiolysis only with benzodiazepines

Exclusion Criteria:

1. Known drug intolerance/allergy: dexmedetomidine or to other ingredients
2. Lacking willingness to save and hand out pseudonymised data within the clinical trial
3. Accommodation in an institution due to an official or judicial order (according to AMG §40 (1) 4)
4. Employee of the Charité - Universitätsmedizin Berlin CVK/CCM
5. Illiteracy
6. Inability to speak and/or read German
7. Minimal mental status examination (MMSE) < 24
8. Severe hearing loss or visual impairment
9. Acute brain injury
10. Intracranial haemorrhage within one year before participation in the study
11. Manifest psychiatric disease
12. Known illicit substance abuse
13. Acute intoxication
14. For women: Pregnancy or positive pregnancy test within the preoperative screening
15. Homeless or other circumstances, where the patient would not be reachable by telephone or postal services for the 3-months follow up
16. Participation in another interventional clinical trial according to the German Drug Law at time of inclusion and during the trial
17. Acute circulatory failure at time of randomisation (severe hypotension with mean arterial pressure < 55 mmHg despite vasopressors or optimal preload)
18. AV-conduction-block II or III (unless pacemaker installed)
19. Severe bradycardia (heart-rate < 50 bpm, preoperative, permanent)
20. Spinal cord injury with known autonomic dysregulation
21. Preoperative acute cerebrovascular event with neurologic residues
22. Liver insufficiency (Child C cirrhosis, MELD Score > 17)
23. Application of Remifentanil during the operation
24. Deep sedation (RASS, -4 to -5)
25. Administration of Clonidine during administration of the study drug
26. Additional administration of Dexmedetomidine within 3 months after study inclusion

Control Group:

Inclusion Criteria:

1. Patients aged ≥ 60 years of European descent (Caucasian)
2. Male or female patients with ASA II+III
3. ASA II+III-patients, for which no operation is planned within the next year
4. No operation in the last half year before study inclusion
5. Offered patient information and written informed consent

Exclusion Criteria

1. Minimal mental status examination (MMSE) < 24
2. Missing informed consent for saving and hand out pseudonymous data
3. Neuropsychiatric morbidity, which limits the conduction of the neurocognitive testing
4. Anacusis or Hypoacusis, which limits the conduction of the neurocognitive testing
5. Taking psychothropic drugs (including sleep-inducing drug and benzodiazepine) on a regular basis and other substances, which limit the conduction of the neurocognitive testing

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2018-03-17 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative delirium | Until the 5th postoperative day
  Incidence of postoperative delirium measured with the Confusion Assessment Method for the ICU (CAM-ICU) or the Confusion Assessment Method (CAM)

SECONDARY OUTCOMES:
Incidence of subsyndromal delirium and severity of postoperative delirium | Until the 14th postoperative day/discharge
  Incidence of Subsyndromal Delirium (SSD) and severity of postoperative Delirium measured with the Intensive Care Delirium Screening Checklist (ICDSC)
Duration of delirium in the intensive care unit | Until the 14th postoperative day/discharge
  Duration of intensive care unit-delirium measured with the Confusion Assessment Method for the ICU (CAM-ICU) and the Intensive Care Delirium Screening Checklist (ICDSC)
Severity of anxiety | Up to three months
  Severity of anxiety measured with the Faces Anxiety Scale (FAS)
Management of sedation | Until the 5th postoperative day
  Management of sedation measured by the Richmond Agitation Sedation Scale (RASS)
Management of vigilance | Until the 5th postoperative day
  Management of Vigilance measured by Glasgow Coma Scale (GCS)
Management of analgesia and pain levels | Up to three months
  Management of analgesia and pain levels measured by Numeric Rating Scale - Visualized (NRS-V), the Faces Pain Scale - Revised (FPS-R), the Behavioral Pain Scale (BPS) or the Behavioral Pain Scale for Non-Intubated (BPS-NI)
Relevant medication | Until the 5th postoperative day
Severity of illness | Up to 14 postoperative days
  Severity of illness measured by Sequential Organ Failure Assessment (SOFA-Score), Simplified Acute Physiology Score (SAPS II) and the Acute Physiology and Chronic Health Evaluation (APACHE II)
Mechanical ventilation/weaning failure | Until the 5th postoperative day
Intraoperative cerebral oxymetry | At time of surgery
Processive Electroencephalography and Electromyography (EEG/EMG) -Data (SedLine®) | At time of surgery
Determination of blood levels | Change from baseline complete blood count performance (Sysmex®) and acetylcholinesterase-analysis at third postoperative day
  Complete blood count performance (Sysmex®) and acetylcholinesterase-analysis
Cortisol-analysis | Up to three months
Organ dysfunctions | Up to three months
Infections | Up to three months
  Infections according to surgical site infections (SSI) and according to the US Centers for Disease Control and Preventions (CDC).
ICU length of stay | Participants will be followed for the duration of intensive care stay, an expected average of 2 days
Hospital length of stay | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  Discharge criteria have to be met according to Post Anaesthetic Discharge Scoring System (PADSS) for monitoring patients discharge.
Quality of life | Up to three months
  Quality of life is measured by EQ-5D (EuroQol Group), a measure generating a single index value for health status with considerable potential for use in health care evaluation
Incidence of postoperative cognitive dysfunction | Up to three months
  Incidence of postoperative cognitive dysfunction (POCD) is measured by Cambridge Neuropsychological Test Automated Battery (CANTAB®) and Mini Mental State Examination (MMSE) including subjective memory feeling (Item 10 of the Geriatric Depression Scale (for already included patients the retrospective follow up by telephone interview)), including limitations in daily activities (EQ-5D)
Mortality | Up to three months
Sleep quality | Up to three months
Photomotor reflex | At time of surgery
Changes of hemodynamic parameters in the intraoperative transesophageal echocardiography | At time of surgery
  Hemodynamic aparemters are measured in patients for elective CABG surgery

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Study Director — Charité-University Medicine (Berlin, Germany)
Locations (1):
- Department of Anesthesiology and Operative Intensive Care Medicine, Campus Charité Mitte and Campus Virchow - Klinikum, Charité- Universitätsmedizin, Berlin, Germany

REFERENCES:
- [Derived] Singh A, Brenna CTA, Broad J, Kaustov L, Choi S. The Effects of Dexmedetomidine on Perioperative Neurocognitive Outcomes After Cardiac Surgery: A Systematic Review and Meta-analysis of Randomized Controlled Trials. Ann Surg. 2022 May 1;275(5):864-871. doi: 10.1097/SLA.0000000000005196. Epub 2021 Aug 27. PMID 35543164